CLINICAL TRIAL: NCT05246319
Title: Evaluation of Preoperative Imaging (CT Scan, DOPA-PET and DOTATOC) in Patients With Small Bowel Neuroendocrine Tumors
Brief Title: Preoperative Imaging in Patients With Small Bowel Neuroendocrine Tumors
Acronym: TEGRELE
Status: Completed | Type: Observational
Sponsor: Laurent BRUNAUD (Other)
Responsible Party: Sponsor-Investigator, Laurent BRUNAUD, PI, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2021PI126
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors; Small Intestinal NET; Lymph Node Metastasis
Keywords: Neuroendocrine Tumors; Small Intestinal NET; Lymph Node Metastasis; Radionuclide Imaging; CT scan
MeSH Terms: conditions — Neuroendocrine Tumors; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with small intestine neuroendocrine tumors: Evaluation of preoperative abdominal imaging in patients who underwent an a resection for neuroendocrine tumors
  Interventions: Diagnostic Test: preoperative imaging

INTERVENTIONS:
Diagnostic Test: preoperative imaging — evaluation of preoperative imaging (versus nodes observed on pathology)

SUMMARY:
Digestive NETs are the second most common malignant digestive tumor after adenocarcinoma. The most common gastrointestinal NETs arise from the small intestine. These tumors have a high lymph node and distant metastatic potential (hepatic, pulmonary, etc.). Their management is essentially surgical and the extent of the resection essentially depends on preoperative data from conventional and isotopic imaging.

The goal of surgical resection is to remove the portion of the small intestine carrying the tumour(s) with healthy margins (so-called R0 resection) and affected lymph nodes in the mesentery (lymph node dissection). The extent of lymph node dissection, sometimes significant, exposes you to the risk of short hail with its own complications (malnutrition, diarrhoea, etc.). Consequently, an analysis of the benefits and risks between the interest of an extensive and oncological resection (R0) and the risks of short bowel must be carried out for each patient.

The reference examination to define lymph node involvement is determined by the histological examination of the resected surgical specimen (reference examination). The preoperative evaluation of lymph node extension is done by preoperative abdominal CT scan. However, the preoperative CT scan is not always consistent (sensitivity and specificity) with the pathology data (reference examination). For about 5 years, isotopic imaging (DOPA-PET and DOTATOC) has become feasible and could improve the quality of preoperative evaluation of lymph node extension. Consequently, the aim of this study is to determine the contribution of isotopic imaging (DOPA-PET and DOTATOC) in the preoperative evaluation of lymph node extension.

DETAILED DESCRIPTION:
Digestive neuroendocrine tumors (NET) are developed from neuroendocrine cells, of epithelial origin, scattered throughout the digestive tract. These tumors form a heterogeneous group defined according to the site of origin, the cell type affected, the functional character or not, the cell differentiation (morphology), and finally the potential for tumor progression and aggressiveness. Digestive NETs are the second most common malignant digestive tumor after adenocarcinoma. The most common gastrointestinal NETs arise from the small intestine. These tumors have a high lymph node and distant metastatic potential (hepatic, pulmonary, etc.). Their management is essentially surgical and the extent of the resection essentially depends on preoperative data from conventional and isotopic imaging. The goal of surgical resection is to remove the portion of the small intestine carrying the tumour(s) with healthy margins (so-called R0 resection) and affected lymph nodes in the mesentery (lymph node dissection). The extent of lymph node dissection, sometimes significant, exposes you to the risk of short hail with its own complications (malnutrition, diarrhoea, etc.). Consequently, an analysis of the benefits and risks between the interest of an extensive and oncological resection (R0) and the risks of short bowel must be carried out for each patient.

The reference examination to define lymph node involvement is determined by the histological examination of the resected surgical specimen (reference examination). The preoperative evaluation of lymph node extension is done by preoperative abdominal CT scan. However, the preoperative CT scan is not always consistent (sensitivity and specificity) with the pathology data (reference examination). For about 5 years, isotopic imaging (DOPA-PET and DOTATOC) has become feasible and could improve the quality of preoperative evaluation of lymph node extension. Consequently, the aim of this study is to determine the contribution of isotopic imaging (DOPA-PET and DOTATOC) in the preoperative evaluation of lymph node extension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuroendocrine tumors who underwent a scheduled surgical procedure for small bowel resection

Exclusion Criteria:

* patients without preoperative CT scan
* patients with abdominal resection performed in emergency

Ages: 16 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with neuroendocrine tumors who underwent a scheduled surgical procedure for small bowel resection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
mesenteric lymph nodes | before surgical procedure
  Evaluate the number and location of affected mesenteric lymph nodes (defined by the pathology reference) which were visualized preoperatively by conventional imaging (CT) and isotopic imaging (DOPA-TEP and DOTATOC).

SECONDARY OUTCOMES:
comparison | before surgical procedure
  Compare conventional imaging (CT) and isotopic imaging (DOPA-TEP and DOTATOC) in terms of positive predictive value of nodal involvement

CONTACTS AND LOCATIONS:
Overall Officials: laurent Brunaud, MD, PhD, Principal Investigator — CHRU Nancy
Locations (2):
- France (2):
  - CHRU Nancy, Nancy
  - CHRU Nancy - Département Chirurgie Viscérale, Métabolique et Cancérologique CVMC (7ème étage), Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deguelte S, Hammoutene C, Poncet G, Brunaud L, Perrier M, Kianmanesh R, Cadiot G. Concept of reintervention with thorough lymphadenectomy after suboptimal resection of small-intestine neuroendocrine neoplasms: A multicentre preliminary study. J Neuroendocrinol. 2022 Jun;34(6):e13117. doi: 10.1111/jne.13117. Epub 2022 Apr 18. PMID 35434838
- [Background] Mocellin S, Nitti D. Gastrointestinal carcinoid: epidemiological and survival evidence from a large population-based study (n = 25 531). Ann Oncol. 2013 Dec;24(12):3040-4. doi: 10.1093/annonc/mdt377. Epub 2013 Sep 19. PMID 24050954
- [Background] Dasari A, Shen C, Halperin D, Zhao B, Zhou S, Xu Y, Shih T, Yao JC. Trends in the Incidence, Prevalence, and Survival Outcomes in Patients With Neuroendocrine Tumors in the United States. JAMA Oncol. 2017 Oct 1;3(10):1335-1342. doi: 10.1001/jamaoncol.2017.0589. PMID 28448665
- [Background] Keck KJ, Maxwell JE, Utria AF, Bellizzi AM, Dillon JS, O'Dorisio TM, Howe JR. The Distal Predilection of Small Bowel Neuroendocrine Tumors. Ann Surg Oncol. 2018 Oct;25(11):3207-3213. doi: 10.1245/s10434-018-6676-2. Epub 2018 Jul 27. PMID 30054825
- [Background] Moertel CG. Karnofsky memorial lecture. An odyssey in the land of small tumors. J Clin Oncol. 1987 Oct;5(10):1502-22. doi: 10.1200/JCO.1987.5.10.1502. No abstract available. PMID 2443618